CLINICAL TRIAL: NCT00443183
Title: Emergency Physician Brief Interventions for Alcohol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9906010726; 5R01AA012417-03 (NIH)
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2016-08

CONDITIONS: Harmful Drinking; Hazardous Drinking

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Brief Negotiation Interview (Experimental): The Brief Negotiation Interview is a manual guided intervention using techniques based on motivational interviewing, brief advice, and behavioral contracting and is designed to be delivered in less than 10 minutes.
  Interventions: Behavioral: Brief Negotiation Interview (BNI)
- Discharge Instructions (Placebo Comparator): Scripted discharge instructions to be read by emergency practitioner and designed to be less than 1 minute in length.
  Interventions: Behavioral: Discharge Instructions

INTERVENTIONS:
Behavioral: Brief Negotiation Interview (BNI) — The Brief Negotiation Interview is a manual guided intervention using techniques based on motivational interviewing, brief advice, and behavioral contracting and is designed to be delivered in less than 10 minutes.
  Arms: Brief Negotiation Interview
Behavioral: Discharge Instructions — Used as a placebo comparator, scripted discharge instructions are to be read by emergency practitioner and designed to be less than 1 minute in length.
  Arms: Discharge Instructions

SUMMARY:
Patients with hazardous and harmful alcohol consumption are at increased risk for adverse health consequences and have frequent visits to the Emergency Department(ED). Despite research that has demonstrated the prevalence of alcohol problems in ED patients, there are limited data on the effectiveness of brief intervention (BI) strategies for patients in this setting. The purpose of the current study is to evaluate the effectiveness of a brief intervention, termed Brief Negotiation Interview (BNI), provided by emergency practitioners (EPs-emergency physicians and physician assistants), in reducing alcohol consumption in ED patients with hazardous and harmful drinking. In a controlled randomized clinical trial of 500 patients with hazardous and harmful drinking, BNI will be compared to scripted discharge instructions (DI). Three hypotheses will be tested: BNI is superior to DI in: 1) reducing alcohol consumption; 2) reducing the number of binge drinking episodes; and 3) increasing utilization of primary care or alcohol-related services. Alcohol consumption and utilization of primary care or alcohol-related services will be measured by self-report at 1,6 and 12 months. An additional benefit to changing patterns of consumption and utilization of health services may be decreased ED visits and alcohol-related hospitalizations. These will be assessed utilizing a statewide database. In order to facilitate real-world application of BNI in the ED, the project will result in a BNI manual for EPs and an adherence and competence scale. Unique features of the current project as compared to earlier studies include: 1)use of a credible control condition; 2) enrollment of a heterogeneous population; 3)use of a manual-guided intervention by existing ED staff; 4)systematic assessment of adherence and competence to ensure quality administration and discriminability of interventions; 5)monitoring of use of ancillary treatments; and 6)monitoring of repeat ED visits and alcohol-related hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 18 years or older who present to the adult ED at Yale-New Haven Hospital will be screened for the NIAAA criteria for at risk drinking( ) namely:

  * Men: > 14 drinks per week or > 4 drinks per occasion
  * Women &: > 7 drinks per week or (all >65) > 3 drinks per occasion
  * or will be considered to screen positive for harmful drinking, if they exhibit any current injury or medical condition occurring in the setting of acute alcohol ingestion as determined by a) self-report; b)serum or breathalyzer test with a blood alcohol concentration (BAC) > 0.02mg%;( , , ) or c) a history of any injury or medical condition involving the use of alcohol within the past year.

Exclusion Criteria:

Patients will be excluded for the following:

* Non-English speaking;
* Pregnancy;
* Alcohol dependence;
* Current enrollment in substance abuse treatment program;
* Current cocaine or illicit opiate use;
* Current ED visit for acute psychiatric complaint;
* History of neuroleptic prescription;
* Hospitalization for psychiatric problem in the past year;
* Condition that precludes interview i.e., life threatening injury/illness;
* In police custody; and
* Inability to provide 2 contact numbers for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2002-05; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Number of Drinks Consumed Daily for the Past 30 Days | Baseline (Before Intervention)
Number of Drinks Consumed Per Week | After 6 Months
Number of Drinks Consumed Per Week | After 12 Months
Number of Binge Episodes in the Past 30 Days | After 6 Months
  Greater than 4 drinks for women and greater than 5 drinks for men
Number of Binge Episodes in the Past 30 Days | After 12 Months
  Greater than 4 drinks for women and greater than 5 drinks for men

SECONDARY OUTCOMES:
Contemplation Ladder Scores | After 6 Months
  A brief measure of motivation or readiness to change, allowing patients to indicate their motivation to change their drinking from 1 to 10, in which 2 is least motivated and 10 is most motivated.
Contemplation Ladder Scores | After 12 Months
  A brief measure of motivation or readiness to change, allowing patients to indicate their motivation to change their drinking from 1 to 10, in which 2 is least motivated and 10 is most motivated.
Short Form Health Survey | After 6 Months
  Assess health status in 2 domains, physical and mental, including summary measures and overall general health perceptions.
Short Form Health Survey | After 12 Months
  Assess health status in 2 domains, physical and mental, including summary measures and overall general health perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Gail D'Onofrio, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States